CLINICAL TRIAL: NCT05861752
Title: Paraphilic Disorders and Other Conditions With Risk for Sexual Violence: a Case-control Study
Status: Recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Umeå University (Other)
Responsible Party: Principal Investigator, Josephine Savard, Principal Investigator, Region Stockholm
Other Study IDs: 2022-00430-01
Record Dates: First submitted 2023-05-03; First posted 2023-05-17 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Paraphilic Disorders; Sexual Addiction; Parasomnia
MeSH Terms: conditions — Paraphilic Disorders; Compulsive Sexual Behavior Disorder; Parasomnias | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — We intend to analyze gene variation and epigenetic markers in genes that are related to epigenetic aging and neuroendocrine systems and that may be presumed to have a relationship to aberrant sexual behavior
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical cohort: Patients seeking treatment with Paraphilic disorders, compulsive sexual behavior disorder and/or sexsomnia. These will be explored separately within each condition.
  For procedures, see the Detailed description heading
  Interventions: Behavioral: Treatment as usual
- Healthy controls: Sex- and age-matched controls will be recruited through special research units, and through advertising on e.g. in newspapers, websites and on social media.
  If the person gives written consent, a structured medical assessment is carried out including assessment of psychiatric co-morbidity and medical history.
  The control person will then answer the same questionnaires as the research subjects in the clinical population. They also will be tested regarding impulsivity and provide blood samples.

INTERVENTIONS:
Behavioral: Treatment as usual — both groups will undergo a psychiatric assessment including interviews, impulsivity tests and fill out questionnaires and leave blood samples. The clinical population will be followed regarding treatment as usual
  Groups: Clinical cohort

SUMMARY:
The goal of this case-control study is to compare clinical characteristics in help-seeking individuals with paraphilic disorders or sexsomnia (sexual behaviors during sleep- a diagnosis in the American Psychiatric Association's Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, (DSM-5)), as compared to healthy controls. The main questions this study aims to answer are:

(1a) Is there a difference in experience of violence between the clinical population and healthy controls? Is there a difference between the clinical groups?

(1b) What are the clinical characteristics of these conditions (psychiatric, sociodemographic, and genetic/epigenetic factors)? Does the clinical population differ from healthy controls?

(1c) How are the psychometric properties of the assessment forms (primarily those addressing sexual deviance and compulsive sexuality) in the project?

(1d) How has sexual interest developed over time among patients with paraphilic disorders? (including the person's own description of e.g. triggers and expectations).

Follow-up of clinical population:

(2) What is the typical treatment as usual (TAU) for the patient population? (e.g., average length of care, the percentage of dropouts and what kind of treatment has been given) (3) Are there any factors at baseline (e.g., presence of neuropsychiatric symptoms, age, symptom burden) that predict treatment outcome? (i.e., symptom burden based on self-assessments at follow-up 3, 6 and 12 months from the start of treatment and records in offence registers after 10 years).

DETAILED DESCRIPTION:
After obtaining a written consent, a physician conducts a structured medical assessment including assessment of psychiatric co-morbidity and medical history.

The participant will thereafter answer questions about socio-demographic factors, sexual preference and relational status and answer questionnaires (see last section). Scales that address sleep are used on indication.

Continued assessment include the Mini International Neuropsychiatric Interview (MINI 7.0) and evaluation by a psychologist that focus on the persons sexual behaviour.

The person will also undergo computerized neuropsychological testing of impulsivity and, if consent has been given, also provide a blood samples.

After the assessment phase (intake) we will evaluate psychiatric diagnoses and make a treatment plan.

To answer question 1d (progress description), we will conduct qualitative interviews with 20 persons with sexual deviations. Those participating in this qualitative interview will provide written consent. The interview will take approximately 60 minutes, will be recorded, transcribed, and analyzed qualitatively.

To answer questions 2 and 3, we will after 3, 6 and 12 months note the type of treatment being given (e.g., Cognitive behavioral therapy or pharmacological), the number of completed visits and the number of interrupted treatments.

Treatment is also followed up with questionnaires.

Questionnaires/assessments used in the project:

The Achenbach System of Empirically Based Assessment (ASEBA)

Personality Inventory for DSM-5 (PID-5)

Montgomery Åsberg Depression Rating Scale (MADRS-S)

Hospital Anxiety and Depression Scale (HADS)

Ritvo Autism and Asperger Diagnostic Scale - Screening Tool (RAADS-14).

The Adult ADHD Self-Report Scale - Screen (ASRS-v1.1 Part A).

The Alcohol Use Disorders Identification Test (AUDIT)

The Drug Use Disorders Identification Test (DUDIT).

Childhood Trauma Questionnaire - Short Form (CTQ-SF)

Barratt Impulsiveness Scale (BIS).

The Brief version of the Difficulties in emotional regulation scale (DERS-16)

Brunnsviken Brief Quality of Life Inventory (BBQ)

Revised University of California (UCLA) Loneliness Scale (RULS)

Perceived Social Support (PSS-14)

Perceived Stress Scale (PSS)

Karolinska Interpersonal Violence Scale (KIVS)

Hypersexual Disorder Current assessment scale (HD:CAS)

Compulsive sexual behavior disorder scale (CSBD-19)

Rape scale

Hypersexual Behavior Inventory (HBI)

Client Satisfaction Questionnaire (CSQ-8)

Susceptibility to Temptation Scale (STS)

Långström Self-assessment of Sexual Interests (LASSIE)

Insomnia Severity Index (ISI)

Karolinska sleep questionnaire (KSQ)

Frotteuristic Disorder: Current Assessment Scale (FD: CAS) Voyeuristic Disorder: Current Assessment Scale (VD: CAS) Exhibitionistic Disorder: Current Assessment Scale (ED: CAS) Coercive Sexual Sadism Disorder: Current Assessment Scale (CSSD: CAS)

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and older
2. Signed informed consent
3. Be able to understand the Swedish language in oral and in writing
4. Meet criteria for paraphilia (sexual deviation) according to DSM-5 (with the exception of pedophilia), compulsive sexual behavior disorder according to the International Classification of Diseases (ICD-11), or sexsomnia (sexual act during sleep)

Exclusion Criteria:

1. Serious mental disorder such as current psychosis or severe depression that requires immediate handling/treatment.
2. Psychological condition that may endanger the patient's health or the scientific parts of the study, this is assessed by the assessing physician and psychologist (for example, intellectual disability).

Criteria for control persons:

Inclusion criteria

1. Age and sex matched to clinical population
2. Signed informed consent
3. Be able to understand the Swedish language in oral and in writing

Exclusion criteria

1. Serious somatic illness (determined by the study physician).
2. Ongoing substance use syndrome
3. Serious psychiatric illnesses/conditions that require medical attention (determined by the study physician).
4. First-degree relative with schizophrenia, bipolar disorder or deceased by suicide.
5. Positive screening for compulsive sexual behavior disorder, paraphilia or sexsomnia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinical population: persons seeking treatment at the ANOVA clinic with indication of paraphilic disorder, Compulsive sexual behavior disorder or sexsomnia
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2027-10-19 (Estimated); Study Completion 2037-10-19 (Estimated)

PRIMARY OUTCOMES:
Karolinska interpersonal violence scale | Baseline
  the outcome measure for main question (1a) is the Karolinska interpersonal violence scale (KIVS) that measures exposure to and use of violence. The Karolinska Interpersonal Violence Scale contains 4 rating scales assessing exposure to violence and expressed violent behavior in childhood (between 6-14 years of age) and during adult life (15 years or older). The subscales are scored 0-5. (Min = 0, Max= 20). Higher scores indicate more experience of violence.

SECONDARY OUTCOMES:
The Mini International Neuropsychiatric interview (MINI) | At baseline.
  a validated diagnostic structured interview to assess for mental disorders
Långström Self-assessment Sexual Interests (LASSIE) | At baseline.
  A self-assessment scale based on the diagnostic criteria for paraphilic disorders listed in Screening for paraphilic disorders in the DSM-5
Personality Inventory for DSM-5 (PID-5) | At baseline.
  is a self-assessment of personality-related traits and problems in different domains.
Achenbach System of Empirically Based Assessment | At baseline.
  a self-report questionnaire for adults screening for e.g., behavioural problems. Each item is not directly correlated with a specific scale, instead the assessments recognize patterns of syndromes.
Hypersexual Disorder: Current Assessment Scale (HD:CAS) | At baseline, and after 3, 6 and 12 months for each individual.
  Symptoms of hypersexual disorder. Score range is 0-24. A higher score indicates more severe problems.
The Montgomery-Åsberg Depression Rating Scale - Self rating (MADRS-S) | At baseline, and after 3, 6 and 12 months for each individual.
  Score range is 0-54. A higher score indicates more severe problems.
The Hospital Anxiety and Depression Scale (HADS) | At baseline, and after 3, 6 and 12 months for each individual.
  Score range is 0-21. A higher score indicates more severe problems.
The Barratt Impulsiveness Scale (BIS) | At baseline.
  Score range is 30-120. A higher score indicates more severe problems.
Compulsive Sexual Behavior Disorder Scale-19 (CSBD-19) | At baseline, and after 3, 6 and 12 months for each individual.
  Score range is 19-76. A higher score indicates more severe problems.
The Rape questionnaire (Bumpy 1996). | At baseline, and after 3, 6 and 12 months for each individual.
  Assessment of cognitive distortions about sex. Score range is 36-144. A higher score indicates more severe problems.
Susceptibility to Temptation Scale (STS) | At baseline.
  Score range is 11-55. A higher score indicates more severe problems.
Insomnia Severity Index (ISI) | At baseline, and after 3, 6 and 12 months for each individual with sexsomnia.
  Score range is 0-28. A higher score indicates more severe problems.
The Difficulties in Emotion Regulation Scale (DERS) | At baseline, and after 3, 6 and 12 months for each individual.
  Score range is 16-80. A higher score indicates more severe problems.
Brunnsviken Brief Quality of Life Inventory (BBQ) | At baseline, and after 3, 6 and 12 months for each individual.
  Score range is 0-48. A higher score indicates high quality of life
Client Satisfaction Scale -8 (CSQ-8) | At baseline, and after 3, 6 and 12 months for each individual.
  Score range is 8-32. A higher score indicates higher treatment satisfaction
Revised University of California (UCLA) Loneliness Scale (RULS) | At baseline, and after 3, 6 and 12 months for each individual.
  Score range is 20-80. A higher score indicates more loneliness.
Karolinska Sleep Questionnaire (KSQ) | At baseline, and after 3, 6 and 12 months for each individual with sexsomnia.
  Score range is 13-65. A higher score indicates more severe problems.
DNA/epigenetic markers associated with sexual violence | Collected at baseline.
  Whole blood (DNA-preparation): investigation of NR3C1, NR3C1, FKBP5, CRHR1, CRHR2, LHB, GNRHR, OXTR, CD38, OPRM1, OPRD1, OPRK1, and epigenetic age.
The Hypersexual Behavior Inventory (HBI) | At baseline,and after 3, 6 and 12 months for each individual.
  a 19-item scale constructed to reflect the proposed DSM-5 criteria of hypersexual disorder. Score range is 19-95. A higher score indicates more severe problems.
The Alcohol Use Disorders Identification Test (AUDIT) | At baseline.
  Total score range 0-40, ≥ 8 indicates harmful use.
The Drug Use Disorders Identification Test (DUDIT) | At baseline.
  Total score range 0-44, ≥ 6 indicates harmful use.
The Childhood Trauma Questionnaire - short form (CTQ-SF) | At baseline.
  Consists of 28 items and measures different aspects of childhood abuse and neglect, each with 5 items. Subscale score range: 5-25. A score above 5 indicate experience of trauma/neglect.
Computerized testing of impulsivity Cambridge Gambling Task (CGT) and Stop Signal Task (SST) | At baseline.
  From CANTAB® [Cognitive assessment software]. Cambridge Gambling Task (CGT) Stop Signal Task (SST)
Perceived Stress Scale: (PSS-14) | At baseline.
  Score range is 0-56. A higher score indicates more severe problems.
Perceived Social Support: (PSS) | At baseline, and after 3, 6 and 12 months for each individual.
  Two subscales, one addressing support from family and the other from friends. Score range is 20-80. A higher score indicates more severe problems.
Adult ADHD Self-Report Scale (ASRS) | At baseline.
  A self-report screening scale of adult attention-deficit/hyperactivity disorder (ADHD) consisting of 18 questions about symptoms of adult ADHD. Each item is rated on a 5-point Likert scale with 0="never" and 4="very often". Part A (items 1-6) has four items of inattention and two items of hyperactivity/impulsivity, and could be used for screening
Ritvo Autism and Asperger Diagnostic Scale - Screening Tool (RAADS-14) | At baseline.
  The scale consists of 14 items and total score range from 0 to 42. A score of 14 indicate need for further assessment.
Frotteuristic Disorder:Current Assessment Scale (FD: CAS), Voyeuristic Disorder: Current Assessment Scale (VD: CAS), Exhibitionistic Disorder: Current Assessment Scale (ED: CAS), Coercive Sexual Sadism Disorder: Current Assessment Scale (CSSD: CAS) | At baseline and after 3, 6 and 12 months for each individual. (For research question 1c: within 6 years)
  The questionnaires are all scored 0-32. A higher score indicates more severe problems.
Qualitative interview (Research question 1d) | within 6 years
  A 60 min interview focusing on the disorder progress from first memory to current state.
Description of treatment as usual (Research question 2) | Registration at baseline and after 3, 6 and 12 months for each individual
  Registration if the participant is receiving cognitive behavioral therapy, pharmacological, psychoeducation, number of fulfilled treatments, average treatment duration.
Sociodemographic factors | At baseline (part of clinical evaluation)
  Age, education level, country of origin, gender identity, relationship status, residence, living condition, offspring, employment, sexual orientation, medical treatment
Conviction of sexual offence (Research question 3) | After 10 years
  Convictions in the Swedish offence register

CONTACTS AND LOCATIONS:
Overall Officials: Josephine Savard, MD, PhD, Principal Investigator — Anova, Karolinska University Hospital, Stockholm, Sweden.
Locations (1):
- Josephine Savard, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Individual participants' data that underlie the results of the published article, after deidentification (text, tables, figures and appendices) might be available to researches who provide a methodically sound proposal.